CLINICAL TRIAL: NCT03475732
Title: Pharmacokinetic Study of XueBiJing Injection in Patients With Sepsis
Brief Title: Pharmacokinetics of XueBiJing in Patients With Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Songqiao Liu, Principal Investigator, Southeast University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017ZDSYLL123-P01
Record Dates: First submitted 2018-03-18; First posted 2018-03-23 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Sepsis; Septic Shock; Community Acquired Pneumonia
Keywords: XueBiJing injection; Sepsis; Septic shock; Pharmacokinetics
MeSH Terms: conditions — Sepsis; Shock, Septic; Community-Acquired Pneumonia | interventions — Xuebijing

STUDY DESIGN:
Intervention Model Description: 100mL XueBiJing injection (dissolved with 100 mL of 0.9% normal saline),intravenous infusion for 1.25 h, q12h for 5 days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XueBiJing injection (Experimental): 100mL XueBiJing injection (dissolved with 100 mL of 0.9% normal saline),intravenous infusion for 1.25 h, q12h for 5 days
  Interventions: Drug: XueBiJing injection

INTERVENTIONS:
Drug: XueBiJing injection — 100mL XueBiJing injection (dissolved with 100 mL of 0.9% normal saline),intravenous infusion for 1.25 h, q12h for 5 days
  Other Names: Tianjin Chase Sun Pharmaceutical Co. LTD

SUMMARY:
Pharmacokinetics and disposition of XueBiJing compounds in patients with sepsis

DETAILED DESCRIPTION:
XueBiJing injection, a five-herb combination approved by Chinese FDA in 2004, has been widely used as an add-on therapy in routine sepsis care in Chinese clinics. A comprehensive pharmacokinetic research on this herbal injection has been conducted in healthy human subjects, and the major circulating XueBiJing compounds, as well as their systemic exposure levels and forms and pharmacokinetic characteristics, have been identified. However, it is known that sepsis may induce hepatic, renal and cardiac dysfunction, alter drug metabolizing enzymes and transporters activities, increase capillary permeability, and induce various pathophysiological changes. All these will affect the concentrations at the action sites and pharmacokinetic characteristics of XueBiJing compounds, which contribute to the injection's overall therapeutic action, thus influencing the anti-septic efficacy of the injection. The purpose of this prospective, open label study is to identify the circulating XueBiJing compounds in patients with sepsis after intravenously dosing XueBiJing injection and their systemic exposure forms and levels, pharmacokinetic characteristics, and the associated inter-patient differences of these XueBiJing compounds.

ELIGIBILITY:
Inclusion Criteria:

* 18≤ age ≤70 years old
* Community acquired pneumonia patients who met the Sepsis-3 criteria from Society of Critical Care Medicine (SCCM) /European Society of Intensive Care Medicine (ESICM) with2 ≤SOFA ≤13
* To use XueBiJing injection as an add-on therapy to treat sepsis decided byclinician
* Informed consent obtained

Exclusion Criteria:

* Diagnosis of sepsis for over 48 h
* Pregnant or lactating women
* Patients with a history of anaphylaxis or allergyto XueBiJing or its component herbs
* Patients participated in an investigational clinical trial within 30 days prior to this study
* Patients unable or unsuitable to participate in this study decided by the investigator (i.e., patients whose death are deemed within 48 h or who poorly adhere to the treatment)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-03-18 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of XueBiJing injection compounds | On 1stand 5th day of giving XueBiJing injection: pre-dose, 1.25 h after starting the infusion, and 0.5, 1, 2, 4, and 8 h after terminating the infusion On 2nd to 4th day of giving XueBiJing injection: pre-dose and 1.25 h after starting the infusion
  Plasma concentrations of XueBiJing injection compounds

SECONDARY OUTCOMES:
Accumulative amounts of XueBiJing compounds in urine | On 1st day of giving XueBiJing injection: pre-dose and 0-3.25 and 3.25-12 h after starting the infusion On 5thday of giving XueBiJing injection:0-3.25 and 3.25-12 h after starting the infusion
  Accumulative amounts of XueBiJing compounds in urine

CONTACTS AND LOCATIONS:
Overall Officials: Chuan Li, Doctor, Study Director — Shanghai Institute of Materia Medica, Chinese Academy of Sciences,China
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
Will work on it.

REFERENCES:
- [Background] Li YP, Qiao YJ, Wu ZX, Yao YM, Yu Y, Wu Y. [Effects of Xuebijing injection on high-mobility group box chromosomal protein 1 in septic rats]. Zhongguo Wei Zhong Bing Ji Jiu Yi Xue. 2007 Apr;19(4):239-41. No abstract available. Chinese. PMID 17448282
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Cheng C, Lin JZ, Li L, Yang JL, Jia WW, Huang YH, Du FF, Wang FQ, Li MJ, Li YF, Xu F, Zhang NT, Olaleye OE, Sun Y, Li J, Sun CH, Zhang GP, Li C. Pharmacokinetics and disposition of monoterpene glycosides derived from Paeonia lactiflora roots (Chishao) after intravenous dosing of antiseptic XueBiJing injection in human subjects and rats. Acta Pharmacol Sin. 2016 Apr;37(4):530-44. doi: 10.1038/aps.2015.103. Epub 2016 Feb 1. PMID 26838074
- [Background] Li X, Cheng C, Wang F, Huang Y, Jia W, Olaleye OE, Li M, Li Y, Li C. Pharmacokinetics of catechols in human subjects intravenously receiving XueBiJing injection, an emerging antiseptic herbal medicine. Drug Metab Pharmacokinet. 2016 Feb;31(1):95-98. doi: 10.1016/j.dmpk.2015.10.005. Epub 2015 Nov 4. PMID 26830081
- [Background] Sinnollareddy MG, Roberts MS, Lipman J, Roberts JA. beta-lactam pharmacokinetics and pharmacodynamics in critically ill patients and strategies for dose optimization: a structured review. Clin Exp Pharmacol Physiol. 2012 Jun;39(6):489-96. doi: 10.1111/j.1440-1681.2012.05715.x. PMID 22519600
- [Background] Blot SI, Pea F, Lipman J. The effect of pathophysiology on pharmacokinetics in the critically ill patient--concepts appraised by the example of antimicrobial agents. Adv Drug Deliv Rev. 2014 Nov 20;77:3-11. doi: 10.1016/j.addr.2014.07.006. Epub 2014 Jul 15. PMID 25038549
- [Background] Harvey RD, Morgan ET. Cancer, inflammation, and therapy: effects on cytochrome p450-mediated drug metabolism and implications for novel immunotherapeutic agents. Clin Pharmacol Ther. 2014 Oct;96(4):449-57. doi: 10.1038/clpt.2014.143. Epub 2014 Jul 2. PMID 24987833